CLINICAL TRIAL: NCT05214586
Title: Conservative Treatment of Ingrown Toenail in Stages I or IIa
Brief Title: Conservative Treatment of Ingrown Toenail
Acronym: TOCON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Extremadura (Other)
Collaborators: University of Valencia (Other)
Responsible Party: Principal Investigator, Alfonso Martínez Nova, Professor, Universidad de Extremadura
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOCON
Record Dates: First submitted 2021-12-30; First posted 2022-01-28 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Ingrown Nail; Nails, Abnormal
Keywords: Ingrown toenail; Conservative treatment; Recurrence; Podiatry; Nail remodelling
MeSH Terms: conditions — Nails, Ingrown; Nails, Malformed; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spiculotomy and application of a Gel Nail (Experimental): A nail spicule removal technique will be performed of the edge or nail edges affected by ingrown toenail. After, a gel nail will be applied to remodeling the nail apparatus and avoid damage of the nail in the lateral fold.
  Interventions: Procedure: Follow up of the clinical stage
- Spiculotomy and Nail Re-education with Gauze Bandage (Active Comparator): A nail spicule removal technique will be performed and a cord of gauze bandage between the nail channel and the sheet will be applied. This technique consists in the removal of the portion of the nail sheet that causes ingrown toenail in order to release the soft parts.
  Interventions: Procedure: Follow up of the clinical stage

INTERVENTIONS:
Procedure: Follow up of the clinical stage — Pain, Swelling, Infection, Patient satisfaction and recurrence of the disease will be measured

SUMMARY:
Ingrown toenail has become one of the most prevalent onychopathies and a frequent reason for consultation in podiatry clinics. In the initial stages of the pathology, conservative treatments are the first choice of therapy. The aim was therefore, to analyze and compare the efficacy of the technique of nail re-education with gauze bandage and nail remodelling for the conservative treatment of onychocryptosis in stage I and IIA, A prospective, longitudinal, randomised clinical trial-type analytical study is proposed. A sample of 20 subjects with stage I and IIA onychocryptosis will be selected. Of these, 10 cases were part of the gauze bandage nail re-education group and the remaining 10 cases were part of the nail remodelling group.

ELIGIBILITY:
Inclusion Criteria:

* Ingrown toenail in stage I or IIa (Mozena Classification)

Exclusion Criteria:

* Patients not allowed for clinical follow-up of the evolution of the pathology.
* Patients presented with deforming pathologies
* Pattens had been surgically operated for ingrown toenail

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Recurrence of the disease | 3 months
  Recurrence is defined as a return of the previous symptoms, regrowth of the nail edge, or patient dissatisfaction with the clinical outcome.

SECONDARY OUTCOMES:
Reported pain | Every clinic visit of the patient until 3 months
  Visual analogue scale of pain (0-10)
Infection | Every clinic visit of the patient until 3 months
  Presence of infection symptoms as oozing or built up fluid around the affected area, bleeding, foul smell, overgrowth tissues around the edges of the toenail or abscess filled with puss.
Swelling | Every clinic visit of the patient until 3 months
  Presence of swelling symptoms as pain, redness and hardardening around the affected toenail.
Patient satisfaction | Every clinic visit of the patient until 3 months
  Patient satisfaction survey (0-10)

CONTACTS AND LOCATIONS:
Locations (1):
- Alfonso Martínez Nova, Plasencia, Cáceres, Spain